CLINICAL TRIAL: NCT00802854
Title: Post Marketing Surveillance Study To Observe Safety And Effectiveness Of Eraxis (Registered) Iv.
Brief Title: Post Marketing Surveillance Study To Observe Safety And Efficacy Of Eraxis® IV
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A8851025
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Candidemia; Other Forms of Candida Infections(Intra-abdominal Abscess, Peritonitis)
Keywords: anidulafungin; safety; efficacy
MeSH Terms: conditions — Candidemia; Peritonitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to collect the safety and efficacy data of Eraxis IV (anidulafungin) 100 mg according to Korea Ministry of Food and Drug Safety regulations.

DETAILED DESCRIPTION:
The objective of this study is to determine any problems or questions associated with Eraxis after marketing, with regard to the following clauses under conditions of general clinical practice, in compliance with the regulation "Re-examination Guideline of New Drugs".

1. Serious adverse event/adverse drug reaction
2. Unexpected adverse event/adverse drug reaction that have not been reflected in the approved drug label.
3. Known adverse drug reaction
4. Non-serious adverse drug reaction
5. Other safety and effectiveness information Eraxis was first approved as a new medicine on 30 May 2008. As required for any new medication approved by Ministry of Food and Drug Safety (MFDS), information on safety and effectiveness of new medication should be researched on certain number of subjects taking the drug in the setting of routine practice during the initial 6 years after the approval of new drug(until 29 May 2014).

However, minimal required number of subjects was not met during the original reexamination period (30 May 2008 ~ 29 May 2014). Therefore, according to an order from MFDS on 02 Mar 2015, Eraxis PMS was requested to collect the rest of required subjects by 02 September 2016 in prospective and retrospective approach.

ELIGIBILITY:
1. Prospective Study Population 1.1. Inclusion Criteria

   Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:
   * Use in the treatment of invasive candidiasis in adult patients
   * Evidence of a personally signed and dated data privacy statement indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

   1.2. Exclusion Criteria

   Subjects presenting with any of the following will not be included in the study:
   * Subjects to whom Eraxis IV is prescribed for other diseases than invasive candidiasis in adult patients.
   * Subjects less than 18 ages should be excluded in this study since safety and effectiveness in pediatric patients have not been established yet.
   * Hypersensitivity to the active substance, or to any of the excipients.
   * Hypersensitivity to other medicinal products of the echinocandin class (e.g. caspofungin).
2. Retrospective Study Population 2.1. Inclusion Criteria

Subjects must meet one of the following inclusion criteria to be eligible for enrollment into the study:

Since all subjects enrolled should meet the usual prescribing criteria as per the local product document of Eraxis IV at the time of starting Eraxis IV administration, the inclusion criteria is divided as followings on the basis of 10 Mar 2015 when the approved indication was updated.

* In case where the starting date of Eraxis IV administration is prior to 10 Mar 2015 - Use in the treatment of the following fungal infections: candidemia and other forms of Candida infections (intra-abdominal abscess, and peritonitis)
* In case where the starting date of Eraxis IV administration is 10 Mar 2015 or after - Use in the treatment of invasive candidiasis in adult patients 2.2. Exclusion Criteria

Subjects presenting with any of the following will not be included in the study:

* Subjects to whom Eraxis IV was prescribed for other diseases than candidemia and other forms of Candida infections (intra-abdominal abscess, and peritonitis) (in case where the starting date of Eraxis IV administration is prior to 10 Mar 2015) or invasive candidiasis in adult patients (in case where the starting date of Eraxis IV administration is 10 Mar 2015 or after).
* Subjects less than 18 ages should be excluded in this study since safety and effectiveness in pediatric patients have not been established yet.
* Hypersensitivity to the active substance, or to any of the excipients.
* Hypersensitivity to other medicinal products of the echinocandin class (e.g. caspofungin).
* Subjects enrolled in the prospective phase study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 subjects will be studied according to the review result by the MFDS for the request for the adjustment of number of subjects.
  To achieve the target sample size, the study is being conducted in prospective study design and retrospective study design.
  1. Prospective Study -Subjects will be enrolled by continuous registration method.
  2. Retrospective Study -Physician should enroll patients consecutively who had received at least one dose of Eraxis IV after Eraxis IV approval date (30 May 2008).
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2012-03-02 (Actual); Primary Completion 2016-05-20 (Actual); Study Completion 2016-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- South Korea (10):
  - Chonbuk National University Hospital, Deokjin-gu, Jeollabuk-do
  - Dong-A University Hospital, Busan
  - Dong-A University Medical Center (Dong-A University Hospital), Busen
  - Keimyung University Dongsan Medical Center (KUDMC), Daegu
  - Daegu fatima hospital, Daegu
  - Daegu Catholic University Medical Center (DCUMC), Daegu
  - Ajou University Hospital, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Seoul Medical Center, Seoul
  - Asan Medical Center, Seoul

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8851025&StudyName=Post%20Marketing%20Surveillance%20Study%20To%20Observe%20Safety%20And%20Efficacy%20Of%20Eraxis%AE%20IV

RESULTS

PARTICIPANT FLOW:
Groups:
- Eraxis: Participants who were receiving Eraxis 100 milligram (mg) injection intravenously (IV) according to the approved indication were observed in this study. The dosage recommendations for Eraxis IV were adjusted solely according to medical and therapeutic necessity and the duration of treatment was based on the participant's clinical response.
Period: Overall Study
Arm/Group | Eraxis
Started | 244
Completed | 244
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of Eraxis.
Arm/Group | Eraxis
Number analyzed (Participants) | 244
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 30 years | 6
  30-39 years | 19
  40-49 years | 26
  50-64 years | 84
  Greater than or equal to (>=) 65 years | 109
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107
  Male | 137

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect. Treatment-emergent were events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs.
Time Frame: From the time of first dosing of Eraxis until 28 calendar days after last dose of Eraxis
Population: Safety analysis set included all participants who received at least 1 dose of Eraxis.
Measure: Count of Participants; unit: Participants
Arm/Group | Eraxis
Number analyzed (Participants) | 244
Participants
  AEs | 141
  SAEs | 102

2. Primary Outcome: Number of Participants With Discontinuations From Study Treatment Due to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: From the time of first dosing of Eraxis until 28 calendar days after last dose of Eraxis
Population: Safety analysis set included all participants who received at least 1 dose of Eraxis.
Measure: Count of Participants; unit: Participants
Arm/Group | Eraxis
Number analyzed (Participants) | 244
Participants | 8

3. Primary Outcome: Duration of Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Duration of AE is the total time (in days) from onset of adverse event till the event is resolved in participants who had at least 1 AE.
Time Frame: From the time of first dosing of Eraxis until 28 calendar days after last dose of Eraxis
Population: Subset of safety analysis set which included all participants who had at least 1 AE.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Eraxis
Number analyzed (Participants) | 141
days | 4.03 (5.81)

4. Primary Outcome: Number of Adverse Events (AEs) by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs were classified according to the severity in 3 categories a) mild - AEs does not interfere with participant's usual function b) moderate - AEs interferes to some extent with participant's usual function c) severe - AEs interferes significantly with participant's usual function.
Time Frame: From the time of first dosing of Eraxis until 28 calendar days after last dose of Eraxis
Population: Safety analysis set included all participants who received at least 1 dose of Eraxis.
Measure: Number; unit: events
Arm/Group | Eraxis
Number analyzed (Participants) | 244
events
  Mild | 33
  Moderate | 43
  Severe | 109

5. Primary Outcome: Number of Participants With Outcome in Response to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Outcome of an AE was response to a question answered by those participants who had at least 1 AE: 'Is the adverse event still present?' as 'yes' (when AE was still present), 'unknown' (no information) or 'no, resolved' (when AE was not present and was resolved).
Time Frame: From the time of first dosing of Eraxis until 28 calendar days after last dose of Eraxis
Population: Subset of safety analysis set which included all participants who had at least 1 AE.
Measure: Count of Participants; unit: Participants
Arm/Group | Eraxis
Number analyzed (Participants) | 141
Participants
  Yes | 106
  Unknown | 7
  No, resolved | 28

6. Primary Outcome: Percentage of Treatment-Emergent Treatment-Related Adverse Events (AEs)
Description: AE=any untoward medical occurrence attributed to study drug in participant who received study drug. Treatment-emergent AE=AE between first dose of study drug up to 28 days after last dose that were absent before treatment/worsened relative to pretreatment state. Relatedness of AE to treatment assessed by physician as:Certain=clinically reasonable reaction on cessation of treatment;Probable/likely=followed reasonable time sequence from administration of treatment which was not explained by other drug/chemical substance/accompanying disease;Possible=followed reasonable time sequence from administration of treatment;Unlikely=not likely to have reasonable causal relationship with treatment, seems temporary;Conditional/unclassified=needed more data to make appropriate assessment/its additional data were being reviewed;Unaccessible/unclassifiable=lack of sufficient information hampered accurate causality assessment. % of AEs=(Number of AEs for specified categories/total number of AEs)*100.
Time Frame: From the time of first dosing of Eraxis until 28 calendar days after last dose of Eraxis
Population: Safety analysis set included all participants who received at least 1 dose of Eraxis.
Measure: Number; unit: percentage of AEs
Units Other Than Participants: AEs
Arm/Group | Eraxis
Number analyzed (Participants) | 244
Number analyzed (AEs) | 185
percentage of AEs
  Certain | 1.08
  Probable/likely | 0
  Possible | 5.95
  Unlikely | 92.43
  Conditional/unclassified | 0
  Unaccessible/unclassifiable | 0.54

7. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, red blood cell count, platelet count, white blood cell count, total neutrophils, basophils, lymphocytes); liver function (aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine); electrolytes (sodium, potassium, chloride, calcium, magnesium, phosphate); urinalysis (urine protein). Laboratory abnormalities were identified by the Investigator.
Time Frame: From the time of first dosing of Eraxis until 28 calendar days after last dose of Eraxis
Population: Safety analysis set included all participants who received at least 1 dose of Eraxis. Here, "number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Eraxis
Number analyzed (Participants) | 240
Participants | 35

8. Primary Outcome: Number of Participants With Clinical Response (CR)
Description: CR was categorized as: a) Cure: resolution of signs and symptoms attributed to Candida infection; b) Improvement: significant, but incomplete resolution of signs and symptoms of the Candida infection c) Failure: no significant improvement in signs and symptoms of Candida infection, or death due to the Candida infection; d) Unevaluable: evaluation was not made due to withdrawal of participant from the study prior to assessment of cure or failure, or when lost to follow-up.
Time Frame: From the time of first dosing of Eraxis until 28 calendar days after last dose of Eraxis
Population: Effectiveness analysis set included participants who had been administered Eraxis IV 100 mg at least once and evaluated upon its related effectiveness endpoints at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Eraxis
Number analyzed (Participants) | 199
Participants
  Cure | 88
  Improvement | 89
  Failure | 19
  Unevaluable | 3

9. Primary Outcome: Number of Participants With Mycological Response (MR)
Description: In case cultivation was performed, isolated pathogens before and after administration of Eraxis were recorded and MR outcomes after Eraxis administration were evaluated. MR was evaluated as: a) Eradication: baseline pathogen not isolated from original site culture; b) Presumed eradication: culture data did not exist and CR was defined as cure(resolution of signs and symptoms attributed to Candida infection) or improvement (significant, but incomplete resolution of signs and symptoms of Candida infection); c) Persistence: any baseline Candida species was present in repeat culture; d) Presumed persistence: culture data did not exist and CR was defined as failure (no significant improvement in signs and symptoms of Candida infection, or death due to Candida infection); e) Unevaluable: when culture data did not exist; and f) Superinfection: emergence of new Candida infection at original site of infection or at distant infection site.
Time Frame: From the time of first dosing of Eraxis until 28 calendar days after last dose of Eraxis
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Eraxis
Number analyzed (Participants) | 199
Participants
  Eradication | 149
  Presumed eradication | 28
  Persistence | 16
  Presumed persistence | 6
  Unevaluable | 0
  Superinfection | 0

10. Primary Outcome: Number of Participants With Overall Response (OR)
Description: OR: final effectiveness evaluation analyzed using following criteria (based on physician's evaluation of CR & MR): a)Effective:clinical success (cure/improvement) & microbiological success (eradication/presumed eradication), b)Ineffective:clinical failure/microbiological failure (persistence/presumed persistence); c)Unevaluable:unevaluable CR & MR & neither response was failure. CR:cure (resolutions of symptom), improvement (significant but incomplete resolution of sign/symptom), failure (no significant improvement/death), Unevaluable:no evaluation as participant withdrew prior assessment of cure/failure/lost to follow-up. MR:eradication (baseline pathogen not isolated from original site culture); presumed eradication(culture data not exist & CR of cure/improvement); persistence (baseline Candida species present in repeat culture); presumed persistence (culture data not exist;CR defined as failure), unevaluable:culture data not exist, superinfection:emergence of new Candida infection.
Time Frame: From the time of first dosing of Eraxis until 28 calendar days after last dose of Eraxis
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Eraxis
Number analyzed (Participants) | 199
Participants
  Effective | 173
  Ineffective | 26
  Unevaluable | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Arm/Group | Eraxis
Serious Adverse Events (participants affected / at risk) | 102/244
Other Adverse Events (participants affected / at risk) | 52/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eraxis (N=244)
MULTIPLE ORGAN FAILURE (General disorders) | 7
CARDIAC FAILURE (Cardiac disorders) | 2
SHOCK (Cardiac disorders) | 1
BRAIN HYPOXIA (Nervous system disorders) | 1
MENINGOENCEPHALITIS (Nervous system disorders) | 1
GI HAEMORRHAGE (Gastrointestinal disorders) | 1
CARDIAC ARREST (Cardiac disorders) | 3
FIBRILLATION VENTRICULAR (Cardiac disorders) | 1
TACHYCARDIA VENTRICULAR (Cardiac disorders) | 1
CHOLANGITIS (Hepatobiliary disorders) | 1
COMA HEPATIC (Hepatobiliary disorders) | 1
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 2
ACIDOSIS (Metabolism and nutrition disorders) | 2
ENDOCARDITIS (Vascular disorders) | 2
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
GASTRIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
GI NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
OVARIAN CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PANCREAS NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PULMONARY CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RECTAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
INFECTION BACTERIAL (Infections and infestations) | 1
CANDIDIASIS (Infections and infestations) | 2
PERITONITIS (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 45
CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 8
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY INSUFFICIENCY (Respiratory, thoracic and mediastinal disorders) | 3
RENAL FAILURE ACUTE (Renal and urinary disorders) | 3
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eraxis (N=244)
FEVER (General disorders) | 6
MEDICINE INEFFECTIVE (General disorders) | 2
HYPERTENSION (Cardiac disorders) | 4
HYPOTENSION (Cardiac disorders) | 1
CONVULSIONS (Nervous system disorders) | 3
SPINAL STENOSIS (Nervous system disorders) | 1
ADRENAL INSUFFICIENCY (Endocrine disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
AMYLASE INCREASED (Gastrointestinal disorders) | 1
COLITIS (Gastrointestinal disorders) | 1
COLITIS PSEUDOMEMBRANOUS (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 2
GASTRIC ULCER HAEMORRHAGIC (Gastrointestinal disorders) | 1
GI HAEMORRHAGE (Gastrointestinal disorders) | 1
ILEUS (Gastrointestinal disorders) | 1
MELAENA (Gastrointestinal disorders) | 3
NAUSEA (Gastrointestinal disorders) | 1
FIBRILLATION ATRIAL (Cardiac disorders) | 1
BILIRUBINAEMIA (Hepatobiliary disorders) | 6
GAMMA-GT INCREASED (Hepatobiliary disorders) | 1
SGOT INCREASED (Hepatobiliary disorders) | 2
SGPT INCREASED (Hepatobiliary disorders) | 3
LIPASE INCREASED (Metabolism and nutrition disorders) | 1
PHOSPHATASE ALKALINE INCREASED (Metabolism and nutrition disorders) | 3
DELIRIUM (Psychiatric disorders) | 3
DEPRESSION (Psychiatric disorders) | 1
INSOMNIA (Psychiatric disorders) | 2
ABSCESS (Infections and infestations) | 1
HERPES NOS (General disorders) | 1
INFECTION AGGRAVATED (General disorders) | 1
INFECTION BACTERIAL (Infections and infestations) | 1
INFECTION FUNGAL (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 1
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1
DECUBITUS ULCER (General disorders) | 1
MEDICATION ERROR (General disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 2
SKIN INFECTION (Skin and subcutaneous tissue disorders) | 1
AZOTAEMIA (Renal and urinary disorders) | 1
THROMBOSIS (Vascular disorders) | 1
RETINITIS (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.